CLINICAL TRIAL: NCT05228964
Title: Focused Ultrasound Amygdala Neuromodulation for the Mechanistic Treatment of Affective Disorders
Brief Title: Focused Ultrasound Amygdala Neuromodulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Greg Fonzo, Assistant Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000137
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Depression; Anxiety Disorders; Bipolar Depression; Ptsd
Keywords: amygdala; focused ultrasound; neuromodulation; affective disorder; fMRI
MeSH Terms: conditions — Depression; Anxiety Disorders; Bipolar Disorder; Stress Disorders, Post-Traumatic; Mood Disorders

STUDY DESIGN:
Intervention Model Description: Single arm, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Open-label focused ultrasound (Experimental): Focused ultrasound at a 10 Hz pulse repetition frequency, 5% duty cycle, and 720 mw/cm squared de-rated spatial peak temporal average intensity, delivered over 10 min once a day, five days a week for 3 weeks.
  Interventions: Device: Focused ultrasound

INTERVENTIONS:
Device: Focused ultrasound — Focused ultrasound at a 10 Hz pulse repetition frequency, 5% duty cycle, and 720 mw/cm squared de-rated spatial peak temporal average intensity, delivered over 10 min.

SUMMARY:
The purpose of the study is to examine the feasibility and potential efficacy of low-intensity focused ultrasound as a method of modulating amygdala function to promote improvements in symptoms of an affective disorder. Ultrasound is frequently and safely utilized for diagnostic purposes. In this study, the investigators will utilize magnetic resonance imaging (MRI) and neuronavigation to target the left amygdala and apply ultrasound. This will be conducted once a day, 5 days a week, for 3 weeks. This will be an open-label, single-arm trial.

DETAILED DESCRIPTION:
Affective disorders broadly defined, including the diagnoses of major depression, bipolar disorder, anxiety disorders, and posttraumatic stress disorder, constitute a large portion of the mental health diagnoses worldwide and pose an enormous public health problem. All of these diagnoses are characterized by a common disturbance in affect and emotion, primarily exaggerated and prolonged states of negative affect (e.g., sadness, fear, anxiety, and anger) triggered by reactivity to emotionally provocative stimuli (e.g., a stressful life situation, perceived threat in the environment, etc.). Apropos, all of these diagnoses are similarly characterized by a shared emotion-processing hyperactivity in a subcortical limbic brain structure underlying the detection of salient environmental stimuli-the amygdala. This shared amygdala hyper-reactivity in affective disorders is thought to underlie a common exaggerated emotional reactivity phenotype, consistent with recent conceptualizations of mental illness as reflecting extremes of functioning on trans-diagnostic dimensions of normal bio-behavioral brain processes, i.e. the Research Domain Criteria, which identify the amygdala as a key mediator of all subdomains of negative valence brain systems. Thus, the amygdala remains one of the most promising affective disorder neuromodulatory therapeutic targets.

Although effective psychotherapeutic and pharmacological interventions have been developed for the treatment of affective disorders, a substantial number of individuals fail to respond to such first-line interventions. This inadequacy has led to the development of neuromodulatory therapies for affective disorders, including transcranial electrical (TES)and transcranial magnetic stimulation (TMS), which are believed to exert indirect therapeutic effects on subcortical limbic and ventral prefrontal brain structures via cortical pathways accessible to non-invasive modulation. However, TES/TMS stimulation is critically limited by the fact that focal depth can only reach several centimeters past the skull, thereby limiting the focus of neuromodulation to superficial cortical regions. The investigators propose the inability to directly and non-invasively focally modulate the amygdala, a key locus of affective disorder pathophysiology, is a critical barrier to maximizing the efficacy of neuromodulatory interventions in humans.

Recent advances in brain modulation have identified transcranial low intensity focused ultrasound pulsation (LIFUP) as a novel methodology for reversibly augmenting brain function. LIFUP involves the administration of high frequency sound waves into the brain via a series of transducers placed against the side of the head. This procedure is safe and non-invasive and demonstrates great potential for development as a future neuromodulatory intervention. Importantly, ultrasound has been demonstrated in both animals and humans to have the capability for reversibly up or down-modulating brain function on time scales of seconds to hours.

Crucially, LIFUP has several key advantages over existing non-invasive neuromodulatory interventions. First, it is both focal and depth-compatible, which allows deep subcortical brain structures, e.g., the amygdala, to be directly stimulated non-invasively. Second, it is inherently compatible with functional magnetic resonance imaging (fMRI), the gold-standard methodology for non-invasive brain mapping in humans, which is in contrast to TES/TMS interventions that pose serious risks for deployment in an MR-environment. This allows the modulatory effect of LIFUP to be tracked and quantified in real-time, thereby affording a substantial advancement in stimulation targeting and assessment of target engagement. However, as this technology is very new, there is currently little known regarding its utility as an intervention tool. The investigators will utilize a novel LIFUP device that is capable of directly and non-invasively modulating function of deep subcortical structures such as the amygdala.

In this study, the investigators will test how LIFUP amygdala neuromodulation impacts the function of the amygdala, how this differs in individuals with an affective disorder, and whether repetitive LIFUP targeted to the amygdala (5 days a week for 3 weeks, 15 sessions total) demonstrates any therapeutic benefit on affective disorder symptoms and how such therapeutic benefits might relate to changes observed in brain function.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-65
* Willing and able to undergo the MRI and LIFUP procedures and repeated LIFUP for up to 15 sessions
* English language proficiency sufficient to speak to investigators and understand investigator instruction
* Can visit the laboratory several times over the course of 2 to 6 weeks
* Individuals with a primary affective disorder diagnosis (major depression, bipolar disorder, an anxiety disorder, or posttraumatic stress disorder on the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders Diagnosis 5th Edition
* Score of 19 or greater on the general distress subscale of the 30-item Mood and Anxiety Symptom Questionnaire
* Psychiatric medication(s) on a stable dosage and regimen for the past 3 months (including antidepressants, mood stabilizers, atypical antipsychotics, and sedatives/hypnotics)

Exclusion Criteria:

* Contraindications to LIFUP or MRI including, but not limited to, history of stroke, brain tumors, brain hemorrhages, internal wires, electrodes, pacemakers, implants, irremovable ferromagnetic objects in head that are unsafe for MRI and/or cause large distortions in imaging data, history of seizures (except febrile seizures in childhood), brain surgery, moderate-to-severe head injury or any penetrating head injury, and uncontrolled thyroid disorder.
* Pregnant women or people trying to become pregnant will also be excluded due to the unknown effects of MRI on developing fetuses
* Individuals with serious medical illnesses that are likely to interfere with study: cancer, autism, narcolepsy etc.
* Current active suicidal/homicidal ideation (or suicide attempt in the past 3 months)
* Current substance-use disorder
* Current or recent (within 3 months) psychotic symptoms, or currently meeting diagnostic criteria for a manic episode
* Individuals currently actively engaged in evidence-based or experimental treatments (e.g., weekly cognitive behavioral psychotherapies, transcranial magnetic stimulation, ketamine/esketamine treatment) other than psychiatric medication(s)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on the 30 item Mood and Anxiety Symptom Questionnaire General Distress Subscale score at 6 weeks | Through study completion, around 6 weeks
  A measure of general distress related to mood and anxiety symptoms. Scores range from 10-50, with lower scores indicating less symptoms.
Change from Baseline fMRI activation to emotional stimuli at 6 weeks | Through study completion, around 6 weeks
  Task-based brain activation to emotional faces
Change from Baseline fMRI resting state connectivity at 6 weeks | Through study completion, around 6 weeks
  Connectivity between the left amygdala and the rest of the brain

SECONDARY OUTCOMES:
Change from Baseline Spielberger State-Trait Anxiety Inventory score at 6 weeks | Through study completion, around 6 weeks
  A measure of state and trait anxiety. Scores range from 0 to 60 for each of the sub scales, state anxiety and trait anxiety. Lower scores indicate less anxiety.
Change from Baseline PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders 5th Edition score at 6 weeks | Through study completion, around 6 weeks
  A self-report measure of PTSD symptom severity. Scores range from 0 to 80, with lower scores indicating less PTSD symptoms.
Change from Baseline Snaith Hamilton Pleasure Scale at 6 weeks | Through study completion, around 6 weeks
  A self-report measure of anhedonia. Scoring range from 0 to 14, with lower scores indicating less anhedonia.
Change from Baseline Quick Inventory of Depressive Symptom Self-Report score at 6 weeks | Through study completion, around 6 weeks
  A self report measure of depressive symptoms. Scores range from 0 to 48, with lower scores indicating less symptoms of depression.
Change from Baseline World Health Organization Quality of Life Inventory-Brief subscale scores at 6 weeks | Through study completion, around 6 weeks
  A self-report measure of quality of life with four subscales: Physical Health, Psychological Health, Social Relationships, and Environment. Scores for each range from 4-20, with higher scores indicating better quality of life.
Change from Baseline Beck Depression Inventory II score at 6 weeks. | Through study completion, around 6 weeks
  A self-report measure of depressive symptoms. Scores range from 0 to 63, with lower scores indicating less symptoms of depression.
Change from Baseline Positive and Negative Affect Scale Short Form at 6 weeks. | Through study completion, around 6 weeks.
  A self-report measure of positive and negative affect. There are scores for Positive Affect and Negative Affect, each of which is scored from 10-50. Higher scores indicate more of that particular type of affect.
Change from Baseline Anxiety Sensitivity Index 3 score at 6 weeks | Through study completion, around 6 weeks
  A self-report measure of anxiety sensitivity. Scores range from 0 to 72, with lower scores indicating less anxiety sensitivity.
Change from Beck Anxiety Inventory score at 6 weeks | Through study completion, around 6 weeks.
  A self report measure of anxiety symptoms. Scores range from 0 to 63, with lower scores indicating less anxiety.
Change from Baseline Pittsburgh Sleep Quality Inventory score at 6 weeks | Through study completion, around 6 weeks.
  A self-report measure of sleep quality. Scores range from 0 to 21, with lower scores indicating better quality sleep.
Change from Baseline Temporal Experiences of Pleasure Scale score at 6 weeks. | Through study completion, around 6 weeks.
  A self report measure of hedonic responding. There are two subscales, one assessing anticipatory pleasure and the other assessing consummatory pleasure. Scores for each subscale are the average of the scores for each item on the subscale, ranging from 1 to 6. Higher scores indicate a higher tendency to experience pleasure.
Change from Baseline Urgency-Premeditation-Perseverance-Sensation Seeking-Positive Urgency Short Version score at 6 weeks | Through study completion, around 6 weeks.
  A self-report measure of impulsive behavioral responding. There are 5 subscales, measuring negative urgency, lack of perseverance, lack of premeditation, sensation seeking, and positive urgency. Scores range from 4 to 16, with higher scores indicating greater impulsivity.
Change from Baseline Conor Davidson Resiliency Scale score at 6 weeks | Through study completion, around 6 weeks.
  A self-report measure of resiliency. Scores range from 0 to 40, with higher scores indicating greater resiliency.
Daily Drinking Questionnaire Revised | Through study completion, around 6 weeks
  A self-report measure of daily drinking. Scores range from 0 to no upper bound, as the score reflects the average number of alcoholic drinks consumed over the period assessed.
Change from Baseline Alcohol Use Disorders Identification Test score at 6 weeks | Through study completion, around 6 weeks.
  A self-report measure of problematic alcohol use. Scores range from 0 to 40, with higher scores indicating more problematic alcohol use.
Change from Baseline Cannabis Use Disorders Identification Test score at 6 weeks. | Through study completion, around 6 weeks
  A self-report measure of problematic cannabis use. Scores range from 0 to 32, with higher scores indicating more problematic cannabis use.
Change from Baseline Mood and Anxiety Symptom Questionnaire 30 item Anhedonic Depression subscale score at 6 weeks. | Through study completion, around 6 weeks.
  A subscale measure of anhedonic depressive symptoms. Scores range from 10-50, with lower scores indicating less anhedonic depression.
Change from Baseline Mood and Anxiety Symptom Questionnaire 30 item Anxious Arousal subscale score at 6 weeks. | Through study completion, around 6 weeks
  A subscale measure of anxious arousal symptoms. Scores range from 10-50, with lower scores indicating less anxious arousal.
Change from Baseline Physicians Health Questionnaire 9 score at 6 weeks. | Through study completion, around 6 weeks
  A self-report screener of major depression. Scores range from 0 to 27, with lower scores indicating fewer symptoms of depression.
Change from Baseline Generalized Anxiety Disorder 7 score at 6 weeks. | Through study completion, around 6 weeks
  A self-report screener of generalized anxiety disorder. Scores range from 0 to 21, with lower scores indicating less symptoms of generalized anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Fonzo, Ph.D., Principal Investigator — The University of Texas at Austin
Locations (1):
- Health Discovery Building (HDB), 1601 Trinity St., Bldg B., Z0600, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barksdale BR, Enten L, DeMarco A, Kline R, Doss MK, Nemeroff CB, Fonzo GA. Low-intensity transcranial focused ultrasound amygdala neuromodulation: a double-blind sham-controlled target engagement study and unblinded single-arm clinical trial. Mol Psychiatry. 2025 Oct;30(10):4497-4511. doi: 10.1038/s41380-025-03033-w. Epub 2025 Apr 24. PMID 40275098